CLINICAL TRIAL: NCT00926757
Title: Prophylactic Use of Entecavir for Chemotherapy Associated With Hepatitis B Reactivation in HBsAg (-), Anti-HBc (+) Non-Hodgkin's Lymphoma Patients: a Randomized Controlled Trial
Brief Title: Prophylactic Use of Entecavir for Non-Hodgkin's Lymphoma Patients With Resolved Hepatitis B
Acronym: HBVNHL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, vghtpe user, Yi-Hsiang Huang, Professor, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VGHUST98-P1-07; VGHIRB98-01-08
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Non Hodgkin's Lymphoma; Hepatitis B
Keywords: lymphoma; CD20; Hepatitis B virus; reactivation; Rituximab
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hepatitis B; Lymphoma | interventions — entecavir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Entecavir prophylaxis (Experimental): Participants will initiate entecavir 0.5 mg/day orally on day 1 of the first course of chemotherapy, and will be continued until 3 months after completion of the chemotherapy.
  Interventions: Drug: Entecavir prophylaxis
- Therapeutic arm (Active Comparator): In patients with HBV reactivation and ALT flare > 100 U/L, entecavir 0.5mg daily will be prescribed for the cases till hepatitis remission
  Interventions: Drug: Therapeutic entecavir

INTERVENTIONS:
Drug: Entecavir prophylaxis — Entecavir 0.5mg daily from day 1 of chemotherapy to 3 months after completing chemotherapy
  Other Names: Baraclude
  Arms: Entecavir prophylaxis
Drug: Therapeutic entecavir — Entecavir 0.5cm daily since hepatitis flare and HBV reactivation, till hepatitis remission
  Other Names: Baraclude
  Arms: Therapeutic arm

SUMMARY:
Hepatitis B (HBV) reactivation and hepatitis flare induced by cytotoxic chemotherapy is common in cancer patients who have chronic HBV infection. Lymphoma patients who had previous infected by HBV but negative for HBsAg have a the risk of HBV reactivation during chemotherapy, but prophylactic antiviral treatment is not a routine by current American Association for the Study of Liver Diseases (AASLD) guideline. Prophylactic entecavir might reduce the risk of HBV reactivation in such patients.

DETAILED DESCRIPTION:
Hepatitis B (HBV) reactivation and hepatitis flare induced by cytotoxic chemotherapy is common in cancer patients who have chronic HBV infection. It is best characterized in patients with hematological malignancies such as non-Hodgkin's lymphoma but also can occur in patients with solid tumors. Reactivation during the initiation of chemotherapy may cause delay in cancer treatment and decrease in overall survival. The direct mortality caused by HBV reactivation, predominantly acute liver failure, ranges from 4% to 60%. Based on currently available information, it is well documented that HBV carriers should receive antiviral agents to prevent hepatitis B flare before receiving immunosuppressive agents and chemotherapy. However, development of hepatitis, acute liver failure, and mortality can occur among patients who are HBsAg negative but anti-HBc positive at the time of chemotherapy. Therefore, before the initiation of cytotoxic chemotherapy in cases of non-Hodgkin's lymphoma, it is unknown whether patients previous infected by HBV but negative HBsAg should routinely receive antiviral agents for prevention of HBV flare. In addition, the major concern of long-term lamivudine use is the selection of drug-resistant mutations. Based on these, we designed this current study to address the above important issues. Eligible patients are newly diagnosed, histologically proven anti-CD20-positive non-Hodgkin's lymphoma at our hospital. Patients should be negative of HBsAg but positive of serum anti-HBc. After signing the patient consent form, serum samples will be stored for further genotyping and quantitative HBV DNA testing. Patients will be randomized into two groups. In the prophylactic use group, participants will initiate entecavir 0.5 mg/day orally on day 1 of the first course of chemotherapy. Entecavir treatment will be continued until 3 months after the completion of chemotherapy and achieving the remission of the hepatitis (ALT normalization and undetectable HBV DNA). In the therapeutic use group, patients will start entecavir therapy, 0.5 mg/day orally, only when elevation of ALT (>100 U/L) and HBV DNA (>2000 IU/ml) developed during follow-up, or in the situation of HBsAg reverse seroconversion, and continued entecavir treatment until hepatitis resolved. The primary endpoint is the incidence of HBV reactivation during and within 12 months after completing chemotherapy in diffuse large B cell or follicular lymphoma patients who receive R-CHOP regimen. The secondary endpoint is the incidence of HBsAg reverse seroconversion during and within 12 months after completing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* CD20 positive lymphoma
* negative for HBsAg and positive for anti-HBc
* age over 16 years old
* alanine aminotransferase less than 2 times the upper limit of normal
* bilirubin < 2.5 mg/dL
* neutrophil > 2000/mm3
* platelet > 100,000/mm3
* creatinine < 1.5 mg/dL
* urea nitrogen < 25 mg/dL
* Eastern Cooperative Oncology Group performance score 0 to 2

Exclusion Criteria:

* Child-Pugh class B or C cirrhosis
* grade 2 or greater heart failure by the NYHA classification
* previous chemotherapy,radiotherapy, or concurrent glucocorticoid therapy for other reasons
* other primary liver diseases, such as chronic hepatitis C, hepatitis D, autoimmune hepatitis, or Wilsons' disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the incidence of HBV reactivation during and within 12 months after chemotherapy | Monthly, and till 12 months after chemotherapy

SECONDARY OUTCOMES:
The incidence of HBsAg reverse seroconversion during and within 12 months after completing chemotherapy. | monthly, till 12 months after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hsiang Huang, MD, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital-Division of Gastroenterology, Division of Oncology, Taipei, Taiwan

REFERENCES:
- [Derived] Huang YH, Hsiao LT, Hong YC, Chiou TJ, Yu YB, Gau JP, Liu CY, Yang MH, Tzeng CH, Lee PC, Lin HC, Lee SD. Randomized controlled trial of entecavir prophylaxis for rituximab-associated hepatitis B virus reactivation in patients with lymphoma and resolved hepatitis B. J Clin Oncol. 2013 Aug 1;31(22):2765-72. doi: 10.1200/JCO.2012.48.5938. Epub 2013 Jun 17. PMID 23775967